CLINICAL TRIAL: NCT01159340
Title: Design Compliance Testing of the Icare One Rebound Tonometer According to the American National Standard ANSI Z80.10-2001 and International Standard ISO 8612.2 for Tonometers
Brief Title: Icare Versus Haag-Streit Applanation Tonometer
Status: Completed | Type: Observational
Sponsor: Icare Finland Oy (Industry)
Responsible Party: Markku Eraluoto, CTO, Icare Finland Oy
Other Study IDs: Icare-0021
Record Dates: First submitted 2010-06-30; First posted 2010-07-09 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The clinical performance of Icare ONE Tonometer TA02 was compared to a Goldmann type applanation tonometer (Haag-Streit). Data was collected according to ANSI Z80.10-2003 (ISO 8612.2) standard. Subjects were eligible for the study if they had no exclusion criteria specified in the ANSI/ISO standard. One eye from 260 subjects was selected for the study. The minimum sample size according to the standard is 150. One eye of each subject was selected for the study by an investigator, based on the history of the patient, results of an external examination of the eye with slit lamp, keratometry readings, and prior knowledge of the intraocular pressure (IOP) range. The Icare ONE Tonometer TA02 in comparison to the reference tonometer (Goldmann type tonometer).

ELIGIBILITY:
Inclusion Criteria:

* subjects were eligible for the study if they had no exclusion criteria as specified by the ANSI/ISO standard

Subjects were selected according to the following exclusion criteria (as given in ANSI Z80.10-2003 and ISO 8612):

* subjects with only one functional eye
* those with one eye having poor or eccentric fixation
* high corneal astigmatism (i.e. those eyes displaying an oval contact image with the Goldmann tonometer)
* those with corneal scarring or who have had corneal surgery, including corneal laser surgery
* microphthalmos
* buphthalmos
* contact lens wearers
* dry eyes
* lid squeezers (blepharospasm)
* nystagmus
* keratoconus
* any other corneal or conjunctival pathology or infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were eligible for the study if they had no exclusion criteria specified in the ANSI/ISO standard. One eye from 260 subjects was selected for the study. The minimum sample size according to the ANSI standard is 150. In order to aid enrollment of at least 40 eyes in each pressure range (7-16 mmHg, >16 to <23 mmHg and 23 mmHg or higher), subjects were invited to participate on the basis of prior knowledge of their IOP range. One eye of each subject was selected for the study by an investigator, based on the history of the patient, results of an external examination of the eye with slit lamp, keratometry readings, and prior knowledge of the IOP range.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2009-05; Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Päivi Puska, MD, FEBO, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Glaucoma Service, Department of Opthalmology, Helsinki University Central Hospital, Helsinki, Finland